CLINICAL TRIAL: NCT03865810
Title: Postoperative Outcomes Within an Enhanced Recovery After Surgery Protocol in Gastric Surgery for Cancer (POWER .4)
Brief Title: Postoperative Outcomes Within an Enhanced Recovery After Surgery Protocol in Gastric Surgery for Cancer
Acronym: POWER4
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Responsible Party: Sponsor
Other Study IDs: REDGERM05
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Perioperative Care; Postoperative Complications; Gastric Cancer
MeSH Terms: conditions — Postoperative Complications; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric Surgery: Adult patients undergoing elective gastric surgery for cancer

SUMMARY:
Methods National audit of a 90-day prospective observational cohort in which postoperative complications will be analyzed at 30 days of follow-up in adult patients undergoing scheduled surgery for gastric resection for cancer with or without an intensified recovery program (ERAS : Enhanced Recovery after Surgery) with any level of protocol compliance (from 0-100%)

Research Locations Spanish Hospitals at the state level where these surgical interventions are performed on a regular basis.

Objectives To determine the incidence of postoperative complications per patient and procedure, regardless of the degree of adherence to ERAS protocols and its impact on the hospital stay and postoperative complications including 30-day mortality.

Sample Size For an alpha error of 5% (95% confidence) and an accuracy of 3% and estimating a number of patients with complications of 28%, the sample size calculation yields 861 patients, although the final sample size it may be smaller depending on the proportion of complications detected.

Inclusion criteria Patients older than 18 years who are going to undergo surgery for gastric resection surgery due to cancer regardless of their affiliation to an ERAS intensified recovery program and the compliance level of the protocol (0-100%)

Statistical analysis Continuous variables will be described as mean and standard deviation, if it is a normal distribution, or median and interquartile range, if they are not normally distributed. Comparisons of continuous variables will be performed by one-way ANOVA or the Mann-Whitney test, as appropriate. A univariate analysis will be performed to test the factors associated with postoperative complications, hospital stay and death in the hospital. Univariate analyzes and hierarchical multivariate logistic regression models will be constructed to identify factors associated independently with these results and to adjust for differences in confounding factors. The factors will be introduced in the models based on their relationship with the univariate result (p <0.05), the biological plausibility and the low rate of missing data.

DETAILED DESCRIPTION:
The results of this study will allow to identify, on the one hand, the type of patients presenting postoperative complications and, on the other hand, to identify those items of the ERAS protocols that are independently associated with a reduction in postoperative complications and hospital stay, which will allow to focus the perioperative efforts in those items that actually improve the postoperative outcomes.

Aim 1 will establish the number of patients developing predefined postoperative complications within 30 days of surgery in adult patients undergoing scheduled surgery for gastric resection for cancer with any compliance of an ERAS protocol (including patients with 0 compliance). This will allow us to determine the actual impact of these protocols.

Aim 2 will allow us to know the type of predefined complication presented by the patients included in the ERAS protocols and in patients undergoing colorectal surgery; This will allow, on the one hand, to have a starting point for future clinical trials, and, on the other hand, to focus efforts to avoid these complications.

Aim 3 will allow us to identify those perioperative items of ERAS protocols that are actually associated with a decrease in postoperative complications.

The proposed study will establish a real view of the number of patients presenting postoperative complications that will overcome the limitations of available retrospective studies and provide greater insight into the items of the protocols that are associated with decreased complications; on the other hand, the investigator's hypothesis is that the number of patients who develop predefined postoperative complications within 30 days of surgery decreases as there is greater compliance with the predefined ERAS protocol items

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age undergoing gastric resection surgery due to cancer within or not of an intensified recovery program (ERAS) with any level of compliance with the protocol (from 0-100%).

Exclusion Criteria:

* Patients undergoing emergency surgery

  * Endoscopic procedures
  * Non-oncological gastric surgery
  * Patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age undergoing gastric resection surgery due to cancer
Sampling Method: Non-Probability Sample
Enrollment: 861 (Estimated)
Dates: Start 2019-10-22 (Estimated); Primary Completion 2020-02-22 (Estimated); Study Completion 2020-03-22 (Estimated)

PRIMARY OUTCOMES:
Number of patients with predefined mild-moderate-severe postoperative complications | 30 days after surgery
  Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine were published by the EPCO definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome mesures. infectious complications, cardiovascular complications and other types of complications. Each complication will be graded as mild, moderate or severe.
Number of patients with predefined mild-moderate-severe postoperative complications (gastric cancer surgery specific) | 30 days after surgery
  Each complication will be graded as mild, moderate or severe.

SECONDARY OUTCOMES:
In-hospital all-cause mortality | 30 days after surgery
  The number and percentage of deaths within 30 days of surgery will be reported for each surgical category
Compliance with ERAS items | 30 days after surgery
  Overall compliance will be calculated as the average of all pre- and intraoperative ERAS adapted elements, as specified in the ERAS society colon and rectal guidelines ERAS patients' guideline compliance will be categorised into quartiles
Duration of hospital stay | 30 days after surgery
  The median hospital length of stay (LOS) following the start of surgery, overall, by survival status and by complication status will be reported. Post-operative LOS is the duration in days from the date of the end of surgery to the date of discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ripollés-Melchor, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; Marcos Bruna Esteban, Study Chair — Hospital General Universitario de Valencia, Spain; José M Ramírez Rodríguez, Study Chair — Lozano Blesa University Hospital, Zaragoza, Spain; César Aldecoa, Study Chair — Hospital Universitario Río Hortega, Valladolid Spain; Ane Abad Motos, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; Peter Vorwald, Study Director — Hospital Universitario Fundación Jiménez Díaz. Madrid, Spain; Gloria Crespo, Study Director — Infanta Leonor University Hospital, Madrid, Spain; Carlos Ferrando Ortolá, Study Director — Hospital Clinic of Barcelona; Joaquín Rodríguez Santiago, Study Director — Hospital Mutua Teresa, Spain; José A García Erce, Study Director — Servicio Navarro de Salud - Osasunbidea. Pamplona, Spain
Locations (66):
- Spain (66):
  - Hospital Virgen de los Lirios de Alcoy, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Don Benito-Villanueva de la Serena, Don Benito-Villanueva de La Serena, Badajoz
  - Hospital de Mérida, Mérida, Badajoz
  - Hospital de Igualada, Igualada, Barcelona
  - Hospital Universitario Parc Tauli, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan d'Espi, Barcelona
  - Fundación Hospital del Espíritu Santo, Santa Coloma de Gramanet, Barcelona
  - Hospital Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Vic, Vic, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital General Universitario de Castellón, Castellon, Castellón
  - Hospital Comarcal de Vinaroz, Vinaròs, Castellón
  - Complejo Hospitalario Universitario de A Coruña, A Coruña, Coruña
  - Hospital Universitario Puerta del Mar, Cadiz, Cádiz
  - Complejo Asistencial Universitario de León, León, León
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Getafe, Getafe, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital Comarcal de Inca, Inca, Mallorca
  - Hospital de Manacor, Manacor, Mallorca
  - Hospital Rafael Méndez, Lorca, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Hospital de Manises, Manises, Valencia
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clínic Universitat de Barcelona, Barcelona
  - Hospital Universitario Sant Pau, Barcelona
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario José María Morales Messeguer, Murcia
  - Hospital Reina Sofía, Murcia
  - Complejo Hospitalario y Universitario de Pontevedra, Pontevedra
  - Complejo Hospitalario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Asistencial de Segovia, Segovia
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital Universitario de Álava, Vitoria-Gasteiz
  - Complejo Asistencial de Zamora, Zamora
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ripolles-Melchor J, Abad-Motos A, Bruna-Esteban M, Garcia-Nebreda M, Otero-Martinez I, Abdel-Lah Fernandez O, Tormos-Perez MP, Paseiro-Crespo G, Garcia-Alvarez R, A Mayo-Ossorio M, Zugasti-Echarte O, Nespereira-Garcia P, Gil-Gomez L, Logrono-Ejea M, Risco R, Parreno-Manchado FC, Gil-Trujillo S, Benito C, Jerico C, De-Miguel-Cabrera MI, Ugarte-Sierra B, Barragan-Serrano C, Garcia-Erce JA, Munoz-Hernandez H, Rio-Fernandez SD, Herrero-Bogajo ML, Espinosa-Moreno AM, Concepcion-Martin V, Zorrilla-Vaca A, Vaquero-Perez L, Mojarro I, Llacer-Perez M, Gomez-Viana L, Fernandez-Martin MT, Abad-Gurumeta A, Ferrando-Ortola C, Ramirez-Rodriguez JM, Aldecoa C; POWER Study Investigators Group. Association between use of enhanced recovery after surgery protocols and postoperative complications after gastric surgery for cancer (POWER 4): a nationwide, prospective multicentre study. Cir Esp (Engl Ed). 2023 Oct;101(10):665-677. doi: 10.1016/j.cireng.2023.04.011. Epub 2023 Apr 23. PMID 37094777
- [Derived] Abad-Motos A, Ripolles-Melchor J, Bruna-Esteban M, Ferrando-Ortola C, Paseiro-Crespo G, Abad-Gurumeta A, Garcia-Erce JA, Jerico C, Ramirez JM, Aldecoa C. Postoperative Outcomes Within an Enhanced Recovery after surgery protocol in gastric surgery for cancer (POWER.4): Study protocol for a prospective, multicentre, observational cohort study. Rev Esp Anestesiol Reanim (Engl Ed). 2020 Mar;67(3):130-138. doi: 10.1016/j.redar.2019.10.004. Epub 2019 Nov 22. English, Spanish. PMID 31767197